CLINICAL TRIAL: NCT03889743
Title: Innovative Steroid Treatment to Reduce Asthma Development in Children After First-time Rhinovirus Induced Wheezing - the INSTAR Study
Brief Title: Innovative Steroid Treatment to Reduce Asthma Development in Children After First-time Rhinovirus Induced Wheezing
Acronym: INSTAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Karolinska University Hospital (Other); Haukeland University Hospital (Other); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government); University Hospital of North Norway (Other); Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018/1495; 2024-515350-25-01 (EU CTIS Number)
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Asthma; Inflammation
Keywords: Respiratory Sounds; Steroids; Rhinovirus
MeSH Terms: conditions — Asthma; Inflammation; Respiratory Sounds | interventions — Lactose

STUDY DESIGN:
Intervention Model Description: In Sweden and Finland children who are rhinovirus negative but otherwise fulfill the inclusion criteria, will be included for comparison. They will not be randomized and participate in the intervention but receive follow-up as rhinovirus positive participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone treatment during 3 days
- controls (Placebo Comparator)
  Interventions: Drug: placebo treatment during 3 days

INTERVENTIONS:
Drug: Dexamethasone treatment during 3 days — Dexamethasone 1,0 mg oral tablets. The exact daily dose of dexamethasone will be 0.3 mg/kg (maximum 6.0 mg). The recommended administration of all tablets is to crush the tablets to a smooth powder and then mix with jelly or yogurt. The dissolved dexamethasone is given by mouth and it is recommended to give it in relation to a meal/breastfeeding. If a child vomits within 30 min, the same dose will be given one more time after a break.
  Arms: Dexamethasone
Drug: placebo treatment during 3 days — 1,0 mg oral tablets. The exact daily dose of lactose (instead of dexamethasone) will be 0.3 mg/kg (maximum 6.0 mg). The recommended administration of all tablets is to crush the tablets to a smooth powder and then mix with jelly or yogurt. The dissolved dexamethasone is given by mouth and it is recommended to give it in relation to a meal/breastfeeding. If a child vomits within 30 min, the same dose will be given one more time after a break.
  Other Names: lactose
  Arms: controls

SUMMARY:
The overall objective of the study is to determine the efficacy of corticosteroids in preventing recurrent wheezing and asthma in high-risk, first-time severe wheezing children with rhinovirus infection, stratified by rhinovirus genome load.

The secondary objectives are to determine duration and severity of each acute episode with acute expiratory breathing difficulty, the number of episodes with acute expiratory breathing difficulty, degree of pulmonary hyperreactivity and quality of life within 24 months after study entry.

DETAILED DESCRIPTION:
Asthma is a major and growing public health problem in Norway and beyond. The reason for the increased occurrence of asthma is still poorly understood. However, the disease is a result of a complex interplay between genetic and environmental factors. The current view of asthma pathogenesis is that an abnormal immune response to environmental agents, such as allergens or respiratory viruses, is responsible for initiation and perpetuation of chronic inflammation in genetically susceptible individuals. It is also increasingly evident that asthma originates early in life. However, intervention measures introduced before birth and during the first year of life that reduced or eliminated exposure to house dust, pets, and tobacco smoke together with encouragement of breast-feeding and delayed introduction of solid foods, only had minor effects in preventing asthma development. Thus, there is an urgent need to develop new approaches to asthma prevention in young children.

Recent evidence suggests that rhinovirus infection is a main and independent trigger of acute wheezing and asthma exacerbations in children. Rhinovirus may cause 20-40% of acute wheezing episodes (bronchiolitis) in children during the first 2 years of life, and up to 90% of asthma exacerbations in older children. Rhinovirus etiology of early wheezing is particularly interesting because it has been strongly associated with recurrent wheezing and doctor-diagnosed asthma up to 13 years of age. The strength of this effect has been reported with odds ratios ranging from 3 to 10 during early life. Previously, personal objective markers for increased asthma risk have mainly been related to the presence of atopy development, but atopic disease with eczema generally manifests later, at age 2-3 years. This understanding of early-life rhinovirus associated wheezing as an early marker for asthma has opened a novel opportunity for effective secondary prevention of asthma by identifying children with increased risk of asthma.

Recognizing the role of rhinovirus as an early risk factor for asthma development, has made it essential to control viral effects. Unfortunately, no feasible rhinovirus antivirals are available for children yet.

Rhinovirus infection may lead to broken epithelial barriers facilitating development of inflammation, and asthma is a chronic inflammatory disease of the airways. It is becoming increasingly clear that control of early virus induced inflammation that may develop into chronic inflammation is crucial to intervene with the asthma disease development.

Most cases with bronchiolitis are caused by respiratory syncytial virus (RSV) and rhinovirus. Recent data have shown that RSV is associated with a more severe short-term outcome than rhinovirus, whereas rhinovirus more often than RSV is associated with a more severe long-term outcome related to atopic predisposition and with increased risk of developing asthma. In line with this, several randomized clinical trials (RCT) have failed to show any corticosteroid effect in preventing asthma after early-life infection with RSV. In contrast, and as a major finding that in fact have led to this project, researchers in Turku, Finland have previously reported a post hoc analysis of RCT data showing that a short treatment with oral prednisolone during the first wheezing episode caused by rhinovirus, reduced the risk of recurrent wheezing over the next 1 - 7 years. Moreover, in a prospective single-center RCT, the same researchers confirmed that children with high rhinovirus genome load did benefit from systemic corticosteroids by having fewer recurrences during a 12-month follow-up period and 25% less asthma diagnoses during a 1- and 4-year follow-up.16;17 Hence, asthma after RSV may not be prevented by corticosteroids because RSV infected children less often are atopic and less often develop chronic inflammation, whereas early rhinovirus induced wheezing often occur in genetic predisposed and/or atopic children, and therefore asthma development may be prevented by early corticosteroid intervention. These highly clinically relevant findings must be confirmed in an adequately powered multicenter RCT to fully address the clinical significance of corticosteroid intervention. We expect that this trial will be a landmark in demonstrating long-term disease modifying effects of recurrent wheezing and asthma inception.

ELIGIBILITY:
Inclusion Criteria:

* admitted to pediatric acute wards in the participating hospitals in Norway, Finland, Sweden.
* referred for first severe wheezing episode, defined as first-time acute breathing difficulty with wheezing ever, appearing less than 7 days from onset of symptoms
* one or more of the following:(a) fever, (b) hypoxia (SAT O2 <= 92%), (c) retractions (inter-, subcostal), (d) prolonged expiration (on auscultation), (e) expiratory rhonchi (on auscultation)
* evidence of rhinovirus infection by PCR-test in nasopharyngeal secretions
* signed informed consent and expected cooperation of the patients for the treatment and follow-up must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

* previous episodes with wheezing, defined as a history of acute breathing difficulty with wheezing in need of treatment at a general practitioner or at hospital, or parental information about similar breathing difficulties
* gestational age <37 weeks
* chronic illness other than atopy (eczema),
* previous systemic or inhaled corticosteroid treatment,
* participation to another trial,
* varicella infection or contact during the last 2-3 weeks,
* need for intensive care unit treatment during the present infection, except for respiratory support with non-invasive methods (high flow nasal cannula ventilation, CPAP or BiPAP),
* any reason why, in the opinion of the investigator, the patient should not participate (e.g. not able to comply with study procedures).
* COVID-19 related disease.

Ages: 3 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
time to a new physician-confirmed wheezy episode within 24 months after study entry | 24 months
time to need for a regular controller medication for asthma within 24 months after study entry | 24 months

SECONDARY OUTCOMES:
duration of respiratory symptoms | 24 months
  as determined at the first episode of acute breathing difficulty within 24 months of study entry
severity of respiratory symptoms | 24 months
  as determined at the first episode of acute breathing difficulty within 24 months of study entry
the number of episodes with acute breathing difficulty since start of study medication | 24 months
  as determined at scheduled follow-up visit within 24 months of study entry
the duration of episodes with acute breathing difficulty since start of study medication | 24 months
  as determined at scheduled follow-up visit within 24 months of study entry
the degree of pulmonary hyperreactivity | 24 months
  as determined at scheduled follow-up visit within 24 months of study entry
quality of life: Infant Toddler Quality of Life© (ITQOL©) questionnaire | 24 months
  as determined at scheduled follow-up visit within 24 months of study entry
body height | 24 months
body weight | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Geir Bråthen, Study Director — St. Olavs Hospital
Locations (8):
- Turku University Hospital, Turku, Finland
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Oslo
  - Ullevål University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim
- Karolinska Universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elvebakk T, Dollner H, Partty A, Jartti H, Vuorinen T, Oymar K, Nerheim S, Moe N, Nordbo SA, Follestad T, Koski J, Vollsaeter M, Hofstad A, Klingenberg C, Leknessund CB, Skjerven HO, Risnes K, Soderhall C, Sissener E, Inchley CS, Konradsen JR, Jartti T. INnovative Steroid Treatment to reduce Asthma development in children after first-time Rhinovirus-induced wheezing (INSTAR): protocol for a randomised placebo-controlled trial. BMJ Open. 2025 Jul 30;15(7):e103530. doi: 10.1136/bmjopen-2025-103530. PMID 40738645